CLINICAL TRIAL: NCT03354689
Title: Cervicothoracic Transcutaneous Electrical Nerve Stimulation Attenuates Cardiac Sympathetic Overdrive in Heart Failure: A 123l-MIBG Myocardial Scintigraphy, Randomized Double-Blind Crossover Trial
Brief Title: Transcutaneous Electrical Nerve Stimulation and Cardiac Sympathetic Overdrive in Heart Failure
Status: Completed | Type: Observational
Sponsor: Universidade Federal Fluminense (Other)
Responsible Party: Principal Investigator, Igor Alexandre Fernandes, Post Doctoral Fellow, Universidade Federal Fluminense
Other Study IDs: 39141414.5.0000.5243
Record Dates: First submitted 2017-11-21; First posted 2017-11-28 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Cardiovascular Abnormalities
MeSH Terms: conditions — Cardiovascular Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Scintigraphy — Scintigraphy

SUMMARY:
Introduction: Cardiac sympathetic drive provides inotropic support to the failing heart and preserves cardiovascular homeostasis. Nonetheless, as myocardial insult evolves, this compensatory response leads to a progressive decline in contractile function, increases the vulnerability to arrhythmias and constitutes an independent mortality predictor. Despite advanced pharmacological therapies, side effects and persistent cardiac sympathetic overdrive highlights the modulation of the adrenergic system as a primary target for non-pharmacological strategies in the heart failure (HF) treatment. In this scenario, we will propose cervicothoracic transcutaneous electrical nerve stimulation (TENS) as a non-pharmacological therapy to attenuate cardiac sympathetic overdrive in patients with heart failure. Methods: In this prospective, randomized, sham-controlled, double-blind crossover trial, ten (10) HF patients under optimal pharmacological treatment will be randomly assigned to either an in-home cervicothoracic transcutaneous electrical nerve stimulation therapy (TENS: 30 min twice a day with 80 Hz frequency and pulse duration of 150 μs) or a sham control intervention (SHCI) for two weeks. Following a two-month washout phase from TENS/SHCI, patients crossed over and started the opposite condition. Washout rate and heart-to-mediastinum ratio (planar 123l-metaiodobenzylguanidine myocardial scintigraphy images), indexes of cardiac sympathetic activity and innervation density, muscle sympathetic nerve activity (microneurography) and brachial artery blood flow (Doppler ultrasound) during dynamic handgrip exercise will be obtained at the beginning and end of each condition.

DETAILED DESCRIPTION:
Introduction: Cardiac sympathetic drive provides inotropic support to the failing heart and preserves cardiovascular homeostasis. Nonetheless, as myocardial insult evolves, this compensatory response leads to a progressive decline in contractile function, increases the vulnerability to arrhythmias and constitutes an independent mortality predictor. Despite advanced pharmacological therapies, side effects and persistent cardiac sympathetic overdrive highlights the modulation of the adrenergic system as a primary target for non-pharmacological strategies in the heart failure (HF) treatment. In this scenario, we will propose cervicothoracic transcutaneous electrical nerve stimulation (TENS) as a non-pharmacological therapy to attenuate cardiac sympathetic overdrive in patients with heart failure. Methods: In this prospective, randomized, sham-controlled, double-blind crossover trial, ten (10) HF patients under optimal pharmacological treatment will be randomly assigned to either an in-home cervicothoracic transcutaneous electrical nerve stimulation therapy (TENS: 30 min twice a day with 80 Hz frequency and pulse duration of 150 μs) or a sham control intervention (SHCI) for two weeks. Following a two-month washout phase from TENS/SHCI, patients crossed over and started the opposite condition. Washout rate and heart-to-mediastinum ratio (planar 123l-metaiodobenzylguanidine myocardial scintigraphy images), indexes of cardiac sympathetic activity and innervation density, muscle sympathetic nerve activity (microneurography) and brachial artery blood flow (Doppler ultrasound) during dynamic handgrip exercise will be obtained at the beginning and end of each condition.

ELIGIBILITY:
Inclusion Criteria:

Patients with a diagnosis of heart failure, New York Heart Association (NYHA) functional classification between II to III and left ventricular ejection fraction ≤ 50%

Exclusion Criteria:

* Regular physical activity, pregnancy, unstable angina, acute myocardial infarction in the last 6 months, pacemaker, history of chronic kidney disease (on dialysis) and cardiac surgery.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with heart failure
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2018-09-19 (Actual); Study Completion 2018-10-20 (Actual)

PRIMARY OUTCOMES:
123-MIBG Washout rate | 12 months
  This measurement provides a highly reproducible index of cardiac sympathetic activity
123-MIBG heart-to-mediastinum ratio | 12 months
  This measurement provides a highly reproducible index of cardiac sympathetic innervation
Muscle Sympathetic nerve activity | 12 months
  This measurement provides a highly reproducible index of muscle sympathetic activity

CONTACTS AND LOCATIONS:
Locations (1):
- Fabio A Alves, Niterói, CA, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Campos MO, Nobrega ACL, Miranda SM, Ribeiro ML, Guerra TRB, Braghirolli AMS, Mesquita CT, Fernandes IA. Transcutaneous electrical nerve stimulation attenuates cardiac sympathetic drive in heart failure: a 123MIBG myocardial scintigraphy randomized controlled trial. Am J Physiol Heart Circ Physiol. 2019 Aug 1;317(2):H226-H233. doi: 10.1152/ajpheart.00091.2019. Epub 2019 May 31. PMID 31149841